CLINICAL TRIAL: NCT05839171
Title: Stress Level and the Effect of Mandala Activity Accompanied With Two Different Music on Infertility Women With Embryo Transfer
Brief Title: Mandala Activity Accompanied With Two Different Music on Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, kerime derya beydağ, Assoc. Prof., Istanbul Gedik University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DBEYDAG001*
Record Dates: First submitted 2023-03-30; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Infertility; Stress; Coping Behavior
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Person's Chosen Music + Mandala coloring (Experimental): Every day for at least 20 minutes/7-10 days
  Interventions: Behavioral: music and mandala coloring
- Meditation Music + Mandala coloring (Experimental): Every day for at least 20 minutes/7-10 days
  Interventions: Behavioral: music and mandala coloring
- Standard care (No Intervention): Every day

INTERVENTIONS:
Behavioral: music and mandala coloring — Listening to music and coloring mandalas for women who have undergone embryo transfer and are waiting at home
  Arms: Meditation Music + Mandala coloring; Person's Chosen Music + Mandala coloring

SUMMARY:
In this study; In this study, it is aimed to determine the stress level and the effect of the mandala activity, which is applied to two different musical accompaniments, on coping with stress in infertile women who have undergone embryo transfer.The research was carried out as a randomized controlled experimental study with women who had embryo transfer at Private Samsun Medicana International Hospital IVF Center and Private Samsun VM Medical Park Hospital IVF Center between 01.07.2021 and 31.07.2022. Introductory Information Form, Infertility Stress Scale (PSS), and Infertility Stress Coping Scale (PSSS) were applied to intervention groups with embryo transfer. The intervention group started right after the embryo transfer and performed a mandala activity accompanied by music or meditation music of their own choosing until the day before the BetaHcg test, and the ISS and PSS were repeated one day before the BetaHcg test. Both groups were provided with the application for at least 7-10 days. After embryo transfer to the control group, Introductory Information Form, PSS and PSS were applied, and PSS and PSS were repeated one day before the BetaHCG test, and no intervention was made other than routine practices.

DETAILED DESCRIPTION:
In this study; In this study, it is aimed to determine the stress level and the effect of the mandala activity, which is applied to two different musical accompaniments, on coping with stress in infertile women who have undergone embryo transfer.

The research was carried out as a randomized controlled experimental study with women who had embryo transfer at Private Samsun Medicana International Hospital IVF Center and Private Samsun VM Medical Park Hospital IVF Center between 01.07.2021 and 31.07.2022. Introductory Information Form, Infertility Stress Scale (PSS), and Infertility Stress Coping Scale (PSSS) were applied to intervention groups with embryo transfer. The intervention group started right after the embryo transfer and performed a mandala activity accompanied by music or meditation music of their own choosing until the day before the BetaHcg test, and the ISS and PSS were repeated one day before the BetaHcg test. Both groups were provided with the application for at least 7-10 days. After embryo transfer to the control group, Introductory Information Form, PSS and PSS were applied, and PSS and PSS were repeated one day before the BetaHCG test, and no intervention was made other than routine practices.

ELIGIBILITY:
Inclusion Criteria:

* Being primary infertile,
* Embryo transfer (ET) has been made, Beta Hcg value measurement is in the waiting phase,
* Not receiving psychological counseling from a specialist (psychologist, psychiatrist),
* Mandala activity, yoga, meditation, acupuncture, etc. to relieve stress. not applying a method,
* Not having difficulties in communicating
* Agree to participate in the research.

Exclusion Criteria:

* Being secondary infertile.
* Bleeding, miscarriage, etc. after embryo transfer. to have lived,
* Having difficulties in communicating,
* Applying alternative methods such as mandala activity, yoga, meditation, acupuncture, etc.,
* Receiving psychological counseling from a specialist (psychologist, psychiatrist),
* Not wanting to participate in the research.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women who have undergone embryo transfer and are in the waiting period
Enrollment: 120 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The effect of music and mandala activity on stress level | 8 month
  The COMPI Fertility Problem Stress Scales), The COMPI Fertility Problem Stress Scale, which was validated and reliable in Turkish by Yılmaz , is a 14-item scale that consists of three sub-dimensions and can be applied to both women and men.One of the aims of the study is to reduce the stress level of painting mandala accompanied by music. For this reason, the COMPI scale was filled before the application was made in the first interview with the patients. The patients painted mandala for at least 20 minutes, accompanied by music, every day for 10 days. At the end of the 10th day, the COMPI scale was filled again before the betahcg value was checked.
The effect of music and mandala activity on level of coping with stress | 8 month
  One of the aims of the study is to reduce the stress level of painting mandala accompanied by music. For this reason, the The COMPI Coping Strategy Scales was filled before the application was made in the first interview with the patients. The patients painted mandala for at least 20 minutes, accompanied by music, every day for 10 days. At the end of the 10th day, the The COMPI Coping Strategy Scales was filled again before the betahcg value was checked.

CONTACTS AND LOCATIONS:
Overall Officials: Kerime Derya BEYDAG, Study Director — https://akademik.yok.gov.tr/AkademikArama/view/viewAuthor.jsp
Locations (1):
- Kerime Derya BEYDAG, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van der Vennet, R., & Serice, S. Can Coloring Mandalas Reduce Anxiety? A replication study. Journal of the American Art Therapy Association, 2012,29(2), 87-92.
- [Background] Lee, S. Why Color Mandalas? A Study Of Anxiety-Reducing Mechanisms. Journal of the American Art Therapy Association, 2018,35(1), 35-41.
- [Background] Kim, J., & Kim, S. (2018).The Effect Of Coloring Mandala On Stress and Relaxation In Women Undergoing In Vitro Fertilization Treatment. Journal Of Korean Academy Of Nursing,48(5), 647-655.
- [Background] Maleki, F., Shams, J., & Fallahi Khoshknab, M. (2013). The Effect of Coloring Mandala on Anxiety of Infertile Women. Journal of Caring Sciences, 2(3), 189-195.
- [Background] Ghasemi, M., Dehghani, M., & Tahmasebi, R. (2015). The Effect Of Coloring Mandala On Anxiety And Stress In Infertile Women. International Journal Of Community Based Nursing And Midwifery, 3(3), 214-221.
- [Background] Jafari, Z., & Zarei, E. (2017). The Effect Of Mandala Coloring On The Stress And Anxiety Of Infertile Women. Journal Of Caring Sciences, 6(2), 141-148.
- [Result] Curry, N. A., Kasser, T. Can Coloring Mandalas Reduce Anxiety?. Journal Of The American Art Therapy Association,2005, 22(2), 81-85.